CLINICAL TRIAL: NCT04710498
Title: ML42362: Neoadjuvant Atezolizumab in Surgically Resectable Advanced Cutaneous Squamous Cell Carcinoma
Brief Title: Neoadjuvant Atezolizumab in Surgically Resectable Advanced Cutaneous Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Vasu Divi, Associate Professor of Otolaryngology - Head & Neck Surgery, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-59070; ENT0082 (Other: OnCore)
Record Dates: First submitted 2020-12-09; First posted 2021-01-14 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cutaneous Squamous Cell Carcinoma
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Atezolizumab (Experimental): Subjects will receive neoadjuvant atezolizumab intravenous (IV) infusion at a fixed dose of 1200 mg on Day 1 (+/- 3 days) of each 21-day cycle for a total of 3 doses prior to surgery, unless there is clinical or radiographic evidence of disease progression.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab administered intravenous (IV) infusion at a fixed dose of 1200 mg
  Other Names: RO5541267

SUMMARY:
The purpose of this research is to evaluate whether the administration of atezolizumab before surgical resection of the tumor is feasible and to evaluate the treatment response, safety, and tolerability of atezolizumab.

DETAILED DESCRIPTION:
Primary Objective:

Determine the feasibility of three doses of atezolizumab prior to surgery in patients with advanced cutaneous squamous cell carcinoma

Secondary Objectives:

* Assess response rates to neoadjuvant atezolizumab

  * Objective response rate following completion of neoadjuvant therapy based on RECIST 1.1 criteria
  * Pathological response rate (major and complete pathological response) in final surgical resection specimen
* Assess change in surgical margins or vital structures preserved following neoadjuvant treatment
* Assess safety and tolerability of neoadjuvant atezolizumab

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Age ≥ 18 years at time of signing Informed Consent Form
3. Histologically or cytologically confirmed squamous cell carcinoma
4. Measurable disease per RECIST v1 .1 • Note that protocol specified imaging is not necessary to fulfill this criterion. For example, a patient presenting with a visible 4cm primary lesion who has obviously RECIST evaluable disease may be considered eligible prior to baseline imaging stipulated in the protocol.
5. Availability of a representative tumor specimen that is suitable for determination of PD-L 1 immunohistochemical stain evaluation.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
7. Adequate hematologic and end-organ function appropriate for surgery as determined by routine preoperative evaluation. If liver function, renal function and hematologic laboratory test results are within limits acceptable for elective surgery.

   Laboratory results that will need to be obtained within 28 days prior to initiation of study treatment:

   • Aspartate aminotransferase (AST), Alanine aminotransferas (ALT), total bilirubin, and alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN.).

   • Thyroid-stimulating hormone (TSH) < 13

   • Patients with a history of a high TSH who are receiving levothyroxine replacement at the time of eligibility evaluation and have no clinical evidence of hypothyroidism are eligible.
8. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
9. Negative hepatitis B surface antigen (HBsAg) test at screening
10. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, as defined below: Women must remain abstinent or use contraceptive methods with a failure rate of < 1 % per year during the treatment period and for 5 months after the final dose of atezolizumab. A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state 3 (12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements. Examples of contraceptive methods with a failure rate of< 1 % per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation
11. For men: Agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below: With a female partner of childbearing potential or pregnant female partner, men must agree to remain abstinent or use a condom during the treatment period and for 5 months after the final dose of atezolizumab to avoid exposing the embryo.

Exclusion Criteria:

1. Patients not eligible for standard of care surgical resection
2. Distant metastatic disease
3. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) • Patients with indwelling catheters (e.g., PleurX) are allowed.
4. Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dl or corrected serum calcium > ULN)
5. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis, etc. with the following exceptions: • Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.

   • Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
   * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
   * Rash must cover < 10% of body surface area
   * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
   * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
6. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan History of radiation pneumonitis in the radiation field (fibrosis) is permitted.

7 .Active tuberculosis. Patents do NOT have to be screened for tuberculosis for this trial.

8. Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina

9. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia

10. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment

* Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.

  11. Prior allogeneic stem cell or solid organ transplantation

  12. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications

  13. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab

  14. Current treatment with anti-viral therapy for hepatitis B virus (HBV)

  15. Treatment with investigational therapy within 28 days prior to initiation of study treatment

  16. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti- cytotoxic T-lymphocyteassociated protein 4 (CTLA-4 ), anti-PD-1, and anti-PD-L 1 therapeutic antibodies

  17. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2)) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment

  18. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (TNF)-a agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vasu Divi, MD, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu SS, Colevas AD, Martinez Ramirez L, Megwalu UC, Chen MM, Atwell A, Divi V. Cost of Neoadjuvant Immunotherapy vs Up-Front Surgery in Cutaneous Squamous Cell Carcinoma: A Post Hoc Analysis of a Nonrandomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2025 May 1;151(5):495-502. doi: 10.1001/jamaoto.2025.0001. PMID 40178841

RESULTS

PARTICIPANT FLOW:
Groups:
- Atezolizumab: Subjects received a neoadjuvant atezolizumab intravenous (IV) infusion at a fixed dose of 1200 mg on Day 1 (+/- 3 days) of each 21-day cycle for a total of 3 doses prior to surgery, unless there is clinical or radiographic evidence of disease progression.
  Atezolizumab: Atezolizumab administered intravenous (IV) infusion at a fixed dose of 1200 mg
Period: Overall Study
Arm/Group | Atezolizumab
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Atezolizumab
Number analyzed (Participants) | 20
Age, Customized [Count of Participants; unit: Participants]
  18 to 29 years | 0
  30 to 39 years | 0
  40 to 49 years | 0
  50 to 59 years | 2
  60 to 69 years | 6
  70 to 79 years | 8
  80 to 89 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Complete Neoadjuvant Therapy and Were Eligible for Curative Surgical Resection
Description: Percentage of patients that are able to complete 3 cycles of neoadjuvant atezolizumab and were eligible for curative surgical resection will be measured.
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 20
Participants | 16

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate will be measured based on RECIST v1.1 criteria at baseline, after cycle 2, and at the time or surgery. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of diameters of all target lesions; Progressive Disease (PD), at least a 20% increase in the sum of diameters of target lesions; Overall Response (OR) = CR + PR.
Time Frame: After cycle 3 (duration of each cycle 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 20
Participants
  Complete response | 1
  Partial response | 7
  Stable disease | 10
  Disease progression | 1
  No imaging | 1

3. Secondary Outcome: Pathological Response Rate
Description: Pathological response will be assessed by local pathological review at baseline, after cycle 2, and and at the time or surgery Patients with no viable tumor seen will be classified as a complete pathological response. Patients with < 10% of viable tumor will be classified as a major pathological response.
Time Frame: After cycle 3 (duration of each cycle 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 20
Participants
  Pathological complete response (no viable tumor cells) | 7
  Pathological major response (<= 10% viable tumor cells) | 4
  No pathological response (>10% viable tumor cells) | 8
  No pathological evaluation (surgery declined) | 1

4. Secondary Outcome: Changes in Vital Structures
Description: Assessed changes in vital structures preserved following neoadjuvant treatment
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 19
Participants
  Smaller surgical resection | 10
  Larger surgical resection | 1

5. Secondary Outcome: Changes in Surgical Margins
Description: Assess change in surgical margins preserved following neoadjuvant treatment
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 19
Participants
  Microscopically positive margins | 1
  Microscopically negative margins | 18

6. Secondary Outcome: Safety and Tolerability of Neoadjuvant Atezolizumab
Description: A secondary outcome measure was to assess safety and tolerability of neoadjuvant atezolizumab. Adverse events (AE), serious adverse events (SAE), and treatment-related toxicities were recorded at each study-related visit.
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 20
Participants
  AE's (patients affected) | 20
  SAE's (patients affected) | 1

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=20)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure with Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=20)
Bradycardia (Cardiac disorders) | 1 (1)
Fluid sensation in left ear (Ear and labyrinth disorders) | 1 (1)
Lack of Balance (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Dry Eye (Eye disorders) | 1 (1)
Eye Pain (Eye disorders) | 1 (2)
Eye Pressure (Eye disorders) | 2 (2)
Eyelid Swelling (Eye disorders) | 1 (1)
Periorbital Edema (Eye disorders) | 1 (1)
Facial Pain (General disorders) | 1 (1)
Facial Rash (General disorders) | 2 (2)
Fatigue (General disorders) | 11 (14)
Flu like symptoms (General disorders) | 1 (1)
Lack of Appetite (General disorders) | 2 (2)
Leg pain (General disorders) | 1 (1)
Night Sweats (General disorders) | 1 (1)
Weight Loss (General disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gout (Gastrointestinal disorders) | 1 (1)
Lip Sensitivity (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral Dysesthesia (Gastrointestinal disorders) | 1 (2)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1)
Elevated C-Reactive Protein (Investigations) | 1 (1)
Elevated TSH (Investigations) | 1 (1)
Increased Creatinine (Investigations) | 1 (1)
Increased Total Bilirubin (Investigations) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Nocturnal Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8)
Dizziness, Lightheadedness (Nervous system disorders) | 1 (1)
Facial Nerve Paresis (Nervous system disorders) | 1 (1)
Headache(s) (Nervous system disorders) | 3 (5)
Paresthesia (Nervous system disorders) | 2 (2)
Peripheral Neuropathy (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal/Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cheek Fistula (Skin and subcutaneous tissue disorders) | 1 (1)
Facial Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Fungal Rash/Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT04710498/Prot_SAP_000.pdf